CLINICAL TRIAL: NCT02390323
Title: Changes in Skin Conductance Measurement as an Endpoint Monitor for Sympathetic Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-012
Record Dates: First submitted 2015-02-17; First posted 2015-03-17 (Estimated); Results first posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-07

CONDITIONS: Nerve; Disorder, Sympathetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lumbar Sympathetic Block (Experimental): Patients receiving a Lumbar Sympathetic Block as treatment for lower extremity pain. Skin conductance algesimeter will be used to measure sympathetic activity.
  Interventions: Procedure: Lumbar Sympathetic Block; Device: Skin conductance algesimeter

INTERVENTIONS:
Procedure: Lumbar Sympathetic Block — A lumbar sympathetic block is an injection in the middle of the lower back, toward the left or right side. The "lumbar sympathetic nerves" are a small bundle of nerves that carries "sympathetic" nerve signals from the lower extremities. In some instances, certain injuries to the lower extremities can cause a burning, unusual pain called complex regional pain syndrome or reflex sympathetic dystrophy. Injecting a small amount of local anesthetic on the lumbar sympathetic nerves can identify whether or not this pain is carried by the sympathetic nervous system.
Device: Skin conductance algesimeter — The real-time changes in skin conductance indices can be monitored at the skin level, by use of non-invasive electrodes attached to the skin (similar to EKG electrodes) connected to the skin conductance algesimeter. A computer program analyzes the data and produces a real-time graphic and numeric data demonstrating the skin conductance response. The initiation of successful sympathetic blockade can cause rapid cessation of the skin sympathetic activity that leads to a decrease in skin conductance within seconds.

SUMMARY:
This study is intended to evaluate a monitor that will facilitate ascertainment of an effective sympathetic blockade following Lumbar Sympathetic blocks. Utilization of a monitor with a rapid response and easy clinical applicability which can demonstrate effective sympathetic block would increase efficiency within the procedure suite and also serve to function as an objective endpoint for the evaluation of sympathetic blockade in future research.In current clinical practice, the most commonly used monitoring methods are clinical observations of sympathetic blockade, skin temperature monitoring, pulse pressure monitoring and any combination of these monitoring methods. The skin temperature and pulse pressure may increase after sympathetic block. However, changes in the skin temperature and pulse pressure often demonstrate an unpredictable or delayed response. Confounding variables, such as ambient temperature, coexisting vascular disease, use of other vasoactive medications may contribute to inconsistencies in the temperature or pulse pressure responses.

Normal sympathetic activity stimulates muscarinic receptors in the periphery that subsequently stimulate the sweat glands to secrete and fill with sweat containing sodium and other electrolytes. The electrolytes present in the sweat increase the electrical conductance while decreasing the electrical resistance at the skin level.

The real-time changes in skin conductance indices can be monitored at the skin level, by use of non-invasive electrodes attached to the skin (similar to EKG electrodes). A computer program analyzes the data and produces a real-time graphic and numeric data demonstrating the skin conductance response. The initiation of successful sympathetic blockade can cause rapid cessation of the skin sympathetic activity that leads to a decrease in skin conductance within seconds.

DETAILED DESCRIPTION:
Lumbar sympathetic blocks are clinically used for both diagnosis and treatment of sympathetically mediated pain. in variety of neuropathic pain conditions including complex regional pain syndrome. Sympathetic nerve block has been found successful in about 40% of the patients with neuropathic pain to improve their pain conditions. A sympathetic blockade refers to an injection of a local anesthetic around the sympathetic nerves to alter their functions. The local anesthetic block, often repeated with intervals, may reduce the activity of spontaneous discharges in hyperactive neurons. Reducing the sympathetic nerve activity in the painful region by blocking sympathetic nerve ganglia with a series of local anesthetic nerve blocks may therefore break the cycle of sympathetically mediated pain and provide pain relief. Despite the frequent use of these blocks, there is still a lack of objective methods for determining the successful achievement of sympathetic block in the clinical setting. In current clinical practice, the most commonly used monitoring methods to assess the success of a sympathetic block are observation of clinical signs of sympathetic blockade, skin temperature monitoring, pulse amplitude monitoring in pulse oximetry plethysmography, and any combination of these monitoring methods.

The skin temperature and pulse amplitude in pulse oximetry plethysmography may increase after sympathetic block. However, observation of clinical signs of sympathetic blockade, monitorization of skin temperature, and pulse amplitude often demonstrate an unpredictable or delayed response. Furthermore, confounding variables, such as ambient temperature, coexisting vascular disease, and use of other vasoactive medications, may contribute to inconsistencies in the temperature measurements, or pulse amplitude responses. Therefore, it is a clinical necessity to develop an objective monitoring method that is reliable, rapid response, and also not affected by the other confounders. One potential method is the examination of sympathetic nerve activity via a skin conductance monitor (SCM). Normal skin sympathetic nerve activity stimulates muscarinic receptors that subsequently stimulate the sweat glands to secrete and fill with sweat containing sodium and other electrolytes . The electrolytes present in the sweat increase the electrical conductance while decreasing the electrical resistance at the skin level. The real-time changes in SCM indices can be monitored at the skin level by use of noninvasive electrodes attached to the skin. This is best monitored in the areas with relatively dense sweat glands, such as palm and plantar skin. A computer program analyzes the data and produces real-time graphic and numeric data demonstrating the skin conductance response. The initiation of successful sympathetic blockade can cause rapid cessation of the skin sympathetic nerve activity that leads to a decrease in skin conductance responses within seconds. Currently, there is no rapid response monitor with easy clinical applicability to assess the achievement of a successful sympathetic blockade. Such a monitor could increase procedural accuracy and efficiency, thereby improving patient care. This is especially important in evaluating the response to the sympathetic blocks as they are important for diagnostic purposes to differentiate neuropathic pain types as the sympathetically mediated/maintained pain (SMP), or sympathetically independent pain (SIP). The patients with neuropathic pain presenting with similar symptoms can be classified into two groups depending on their negative or positive response to selective sympathetic blockade. If the pain is relieved by the selective sympathetic block, it is considered SMP. Sympathetically mediated pain is defined as a symptom in a subset of patients with neuropathic pain. The significance of differentiating between SMP or SIP is that SMP has a greater chance of responding favorably to sympatholytic blockade. Therefore, a prospective therapy plan of performing repeated sympatholytic blocks may be considered as these blocks are more efficacious in SMP. On the contrary, as the chance of responding favorably to sympathetic blocks is less likely in SIP, alternative therapies must be considered in this group of patients. In order to plan the prospective treatment options, objective confirmation of sympathectomy created by the attempted sympathetic block is important to differentiate SMP vs SIP. In this context, the utilization of a monitor with a rapid response and easy clinical applicability that can demonstrate effective sympathetic block would serve to function as an objective end point for the evaluation of sympathetic blockade both clinically and for future research. We hypothesize that the SCM is, on average, a more reliable rapid response indicator of a successful sympathetic blockade than traditional monitors such as clinical assessment, monitoring changes in the skin temperature, and pulse amplitude.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for sympathetic block of the lower extremity (lumbar sympathetic block)
* Ages 18-99

Exclusion Criteria:

* Patients with pacemakers or cardiac defibrillators
* Age <18
* IV sedation for anxiolysis or analgesia
* Burn patients or patients with severe dermatologic conditions (as defined by skin conditions causing further pain to patients that actively has to be treated)
* Allergy to adhesive tape
* Patient with diagnosis of: Dysautonomia, Sympathetic dysfunction (e.g.,Raynaud disease, Buerger disease) or Disorders of sweating (e.g.,Acquired idiopathic generalized anhidrosis)
* Patients on vasoactive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Semih Gungor, MD, Principal Investigator — Hospital for Special Surgery, New York

REFERENCES:
- [Background] Storm H. Changes in skin conductance as a tool to monitor nociceptive stimulation and pain. Curr Opin Anaesthesiol. 2008 Dec;21(6):796-804. doi: 10.1097/ACO.0b013e3283183fe4. PMID 18997532

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumbar Sympathetic Block: Patients receiving a Lumbar Sympathetic Block as treatment for lower extremity pain. Skin conductance algesimeter will be used to measure sympathetic activity.
  Lumbar Sympathetic Block: A lumbar sympathetic block is an injection in the middle of the lower back, toward the left or right side. The "lumbar sympathetic nerves" are a small bundle of nerves that carries "sympathetic" nerve signals from the lower extremities. In some instances, certain injuries to the lower extremities can cause a burning, unusual pain called complex regional pain syndrome or reflex sympathetic dystrophy. Injecting a small amount of local anesthetic on the lumbar sympathetic nerves can identify whether or not this pain is carried by the sympathetic nervous system.
  Skin conductance algesimeter: The real-time changes in skin conductance indices can be monitored at the skin level, by use of non-invasive electrodes attached to the skin (similar to EKG electrodes) connected to the skin conductance algesimete
Period: Overall Study
Arm/Group | Lumbar Sympathetic Block
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lumbar Sympathetic Block
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Time to Indication of Successful Blockade Between the Skin Conductance Numeric Value and Bilateral Thermometry.
Description: The skin conductance monitor will be applied immediately prior to the beginning of the procedure. Measurements will be recorded at 0 minutes and every 1 minute until 10 minutes after completion of procedure. Additional measurements will be recorded at the following time points:
  1. Prior to start of procedure (Baseline measurement)
  2. Infiltration of Local Anesthetic
  3. Insertion of the needle
  4. Start of block (First local anesthetic injection after the test dose)
  5. End of block
  6. End of Procedure/Removal of monitor
Time Frame: 10 minutes
Population: Lower back or leg pain
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Lumbar Sympathetic Block
Number analyzed (Participants) | 13
Seconds | 0.08 [.04 to .17]

2. Primary Outcome: Difference in Time to Indication of Successful Blockade Between the Skin Conductance Numeric Value and Unilateral Thermometry.
Time Frame: 10 minutes
Population: Subjects who received a sympathetic nerve block to treat lower back or leg pain
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Lumbar Sympathetic Block
Number analyzed (Participants) | 13
seconds | 0.04 [.01 to .11]

3. Primary Outcome: Hazard Ratio for Time to Successful Blockade Between the Skin Conductance Numeric Value and Plethysmography.
Description: Hazard Ratios are calculated using a Cox proportional Hazards model to compare each traditional method to SCM using a marginal approach with a working independence assumption to account for the correlation between measurements on the same patients. A lower score is a better outcome.
Time Frame: 10 minutes
Population: Lower back or leg pain
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Groups:
- Lumbar Sympathetic Block: Patients receiving a Lumbar Sympathetic Block as treatment for lower extremity pain. Skin conductance algesimeter will be used to measure sympathetic activity.
  Lumbar Sympathetic Block: A lumbar sympathetic block is an injection in the middle of the lower back, toward the left or right side. The "lumbar sympathetic nerves" are a small bundle of nerves that carries "sympathetic" nerve signals from the lower extremities. In some instances, certain injuries to the lower extremities can cause a burning, unusual pain called complex regional pain syndrome or reflex sympathetic dystrophy. Injecting a small amount of local anesthetic on the lumbar sympathetic nerves can identify whether or not this pain is carried by the sympathetic nervous system.
  Skin conductance algesimeter: The real-time changes in skin conductance indices can be monitored at the skin level, by use of non-invasive electrodes attached to the skin (similar to EKG electrodes) connected to the skin conductance algesimeter.
Arm/Group | Lumbar Sympathetic Block
Number analyzed (Participants) | 13
Hazard Ratio | 0.29 [0.14 to 0.63]

4. Primary Outcome: Hazard Ratio for Difference in Time to Indication of Successful Blockade Between the Skin Conductance Numeric Value and Subjective Temperature Difference.
Description: Hazard Ratio for Time to Indication of Successful Blockade Between the Skin Conductance Numeric Value and Subjective Temperature Difference.
  Hazard Ratios are calculated using a Cox proportional Hazards model to compare each traditional method to SCM using a marginal approach with a working independence assumption to account for the correlation between measurements on the same patients. A lower score is a better outcome.
Time Frame: 10 minutes
Population: Subjects who needed a sympathetic nerve block as treatment for lower back or leg pain
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Lumbar Sympathetic Block
Number analyzed (Participants) | 13
Hazard Ratio | 0.06 [0.02 to 0.17]

5. Primary Outcome: Hazard Ratio for Time to Indication of Successful Blockade Between the Skin Conductance Numeric Value and Clinically Visible Hyperemia.
Description: Hazard Ratios are calculated using a Cox proportional Hazards model to compare each traditional method to SCM using a marginal approach with a working independence assumption to account for the correlation between measurements on the same patients.
  The skin conductance monitor will be applied immediately prior to the beginning of the procedure. Measurements will be recorded at 0 minutes and every 1 minute until 10 minutes after completion of procedure. Additional measurements will be recorded at the following time points:
  1. Prior to start of procedure (Baseline measurement)
  2. Infiltration of Local Anesthetic
  3. Insertion of the needle
  4. Start of block (First local anesthetic injection after the test dose)
  5. End of block
  6. End of Procedure/Removal of monitor
  A lower score is a better outcome.
Time Frame: 10 minutes
Population: Subjects who needed a sympathetic nerve block as treatment for lower back or leg pain.
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Lumbar Sympathetic Block
Number analyzed (Participants) | 13
Hazard Ratio | 0.04 [.01 to .13]

6. Primary Outcome: Hazard Ratio for Difference in Time to Indication of Successful Blockade Between the Skin Conductance Numeric Value and Clinically Visible Engorgement of Veins.
Description: as for outcome 5
Time Frame: 10 minutes
Population: Subjects with lower back or leg pain who needed a sympathetic nerve block for its treatment
Measure: Number (95% Confidence Interval); unit: Hazard Ratio
Arm/Group | Lumbar Sympathetic Block
Number analyzed (Participants) | 13
Hazard Ratio | 0.04 [0.01 to 0.13]

ADVERSE EVENTS:
Arm/Group | Lumbar Sympathetic Block
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes